CLINICAL TRIAL: NCT01217034
Title: Phase II Study: Transcatheter Arterial Chemoembolization Therapy In Combination With Sorafenib (TACTICS)
Brief Title: Transcatheter Arterial Chemoembolization Therapy In Combination With Sorafenib
Acronym: TACTICS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kindai University (Other)
Responsible Party: Principal Investigator, Masatoshi Kudo, Professor, Kindai University Faculty of Medicine, Department of Gastroenterology and Hepatology, Kindai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLOG 1001 trial
Record Dates: First submitted 2010-10-02; First posted 2010-10-08 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasm
Keywords: Transcatheter arterial chemoembolization; TACE; sorafenib; Time to untreatable progression; TTUP
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE with sorafenib (Experimental): TACE(on demand) with sorafenib till untreatable progression
  Interventions: Drug: TACE with sorafenib
- TACE alone (Active Comparator): TACE(on demand) till unreatable progression
  Interventions: Procedure: TACE alone

INTERVENTIONS:
Drug: TACE with sorafenib — Sorafenib will be administrated at a dose of 400mg o.d. before the first TACE. After 2days drug rest, TACE will be conducted. Sorafenib will be resumed at a dose of 400mg o.d. from 3 days after TACE(the resumption day can be postponed until 21 days after TACE). When tolerability is confirmed at 1 week after resumption, the dose of sorafenib will be increased to 400mg b.i.d. When tumor increases, TACE will be repeated.
  Other Names: TACE with Nexavar
  Arms: TACE with sorafenib
Procedure: TACE alone — TACE will be conducted at scheduled day. When tumor increases, TACE will be repeated.
  Other Names: TACE
  Arms: TACE alone

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combination therapy with Transcatheter Arterial Chemoembolization (TACE) and sorafenib compared to TACE alone in patients with unresectable hepatocellular carcinoma (HCC) who are not candidates for surgical resection or percutaneous ablation therapy.

DETAILED DESCRIPTION:
TACE with sorafenib Group

Sorafenib will be administrated at a dose of 400mg o.d. before the first TACE. After 2days drug rest, TACE will be conducted. Sorafenib will be resumed at a dose of 400mg o.d. from 3 days after TACE(the resumption day can be postponed until 21 days after TACE). When tolerability is confirmed at 1 week after resumption, the dose of sorafenib will be increased to 400mg b.i.d. When tumor increases, TACE will be repeated.

Control group

TACE will be conducted at scheduled day. When tumor increases, TACE will be repeated.

The treatment regimen will be continued until untreatable progression which is defined as follows:

* Child-Pugh grade C
* Tumor growth (125 percent from baseline status)
* Vascular invasion(Vp3,Vp4)
* Extra hepatic spread which size is more than 10mm

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 Years or over
2. Patients who were fully informed of the study beforehand and signed the informed consent to participate in the study.
3. Patients who are expected to live more than 12 weeks.
4. Patients diagnosed with typical HCC by biopsy,cytology, or diagnostic imaging such as dynamic CT(MRI).Typical HCC is defined by AASLD criteria.
5. Patients in whom complete resection of the tumor by hepatectomy or complete tumor necrosis by local tumor necrosis therapy(RFA) cannot be expected to succeed.
6. Patients with tumors which are confirmed to the liver and can be treated by TACE(the maximum diameter equal to or less than 10cm,and the maximum number of nodule equal to or less than 10).
7. Patients with viable and measurable target lesion.
8. patients with no or one history of TACE therapy.
9. patients with an ECOG PS(Performance Status) Score of 0 or 1.
10. patients with Child-Pugh class A.
11. Patients with laboratory values that meet the following criteria:

    1. Hemoglobin ≥ 8.5 g/dl
    2. Granulocytes ≥ 1500/mm3
    3. Platelet count ≥ 50,000 /mm3
    4. Total serum bilirubin ≤ 3 mg/dl
    5. AST and ALT ≤ 6 times upper limits of normal
    6. Serum creatinine ≤ 1.5 times upper limits of normal

Exclusion Criteria:

1. History of malignant tumor, excluding the following cases:

   1. Curatively treated early stage cancer with a low risk of recurrence ,such as carcinoma in situ of the cervix, basal cell carcinoma, superficial bladder tumor, and early gastric cancer.
   2. Malignant tumor that was curatively treated more than 3 years prior to study entry and has not recurred since then
2. Cardiac disease that meet any of the following criteria:

   1. NYHA Class III or higher congestive heart failure
   2. History of symptomatic coronary artery disease or myocardial infarction within 6 months before enrollment
   3. Arrhythmia requiring control by antiarrhythmic drugs such as beta-blockers or digoxin
3. Serious and active infection, except for HBV and HCV
4. History of HIV infection
5. Renal dialysis
6. Diffuse tumor lesion
7. Extrahepatic metastasis
8. Vascular invasion
9. Intracranial tumor
10. Preexisting or history of hepatic encephalopathy
11. Clinically uncontrolled ascites or pleural effusion
12. Clinically severe gastrointestinal bleeding within 4 weeks of the start of treatment
13. Esophageal and/or gastric varices which has high risk of bleeding
14. History of thrombosis and/or embolism within 6 months of the start of treatment
15. History of receiving any of the following therapies:

    1. Systemic chemotherapy for advanced HCC(including sorafenib therapy)
    2. Local therapy, such as radiofrequency ablation, TACE, or hepatic arterial infusion within 3 months of the start of treatment
    3. Current treatment with CYP3A4 inducing agents
    4. Invasive surgery within 4 weeks of the start of treatment
    5. History of allogenic transplantation
    6. History of bone marrow transplant or haemopoietic stem cell transplant within 4 weeks of the start of this study
16. Unable to take oral medications
17. Gastrointestinal problems that may affect absorption or pharmacokinetics of the study drugs
18. Use of drugs that may affect absorption or pharmacokinetics of the study drugs
19. Concurrent disease or disability that may affect evaluation of the effects of the study drugs
20. Enrollment in another study within 4 weeks of study entry
21. Female patients who are pregnant, lactating, possibly pregnant, or planning to become pregnant
22. Risk of allergic reactions to the study drugs
23. Drug abuse or other physical, psychological , or social problems that may interfere with the participation in the study or evaluation of study results
24. Any condition that could jeopardize the safety of the patient or their compliance in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2010-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | every 8 week
  Patients will be evaluated for these endpoints every 8 weeks
Overall Survival | every 8 week
  The overall survival is defined as time from randomization to death due to any cause, and will be evaluated every 8 weeks in the protocol treatment, and every one year in the follow-up period,respectively.

SECONDARY OUTCOMES:
Time To Progression | every 8 weeks
  Time to progression is defined as time from randomization to radiological progression and will be evaluated every 8 week.
Objective Response Rate | 4week after TACE
  Objective Response Rate is defined as best response
Tumor markers | every 4 weeks
  Change of tumor markers
Safety | every 4 weeks
  Number of participants with adverse events as a measure of safety and tolerability(According to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0)
Time To Untreatable Progression(TTUP) | every 8 week till untreatable progression, assessed up to 100 months
  Time to untreatable progression is defined as time from randomization to untreatable progression and will be evaluated every 8 week.
Time to Child-Pugh C | every 8 week till liver deterioration to Child-Pugh C, assessed up to 100 months
  Time to Child-Pugh C is defined as time from randomization to Child-Pugh C and will be evaluated every 8 week.
Time to intrahepatic tumor progression | every 8 week till intrahepatic tumor progression, assessed up to 100 months
  Time to intrahepatic tumor progression is defined as time from randomization to intrahepatic tumor progression and will be evaluated every 8 week.
Time to vascular invasion | every 8 week till vascular invasion, assessed up to 100 months
  Time to vascular invasion is defined as time from randomization to vascular invasion and will be evaluated every 8 week.
Time to Extrahepatic spread | every 8 week till extrahepatic spread, assessed up to 100 months
  Time to extrahepatic spread is defined as time from randomization to extrahepatic spread and will be evaluated every 8 week.

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Professor, Principal Investigator — Kindai University
Locations (1):
- Kinki University Hospital, Ōsaka-sayama, Osaka, Japan

REFERENCES:
- [Derived] Kudo M, Ueshima K, Ikeda M, Torimura T, Tanabe N, Aikata H, Izumi N, Yamasaki T, Nojiri S, Hino K, Tsumura H, Kuzuya T, Isoda N, Moriguchi M, Aino H, Ido A, Kawabe N, Nakao K, Wada Y, Ogasawara S, Yoshimura K, Okusaka T, Furuse J, Kokudo N, Okita K, Johnson PJ, Arai Y. Final Results of TACTICS: A Randomized, Prospective Trial Comparing Transarterial Chemoembolization Plus Sorafenib to Transarterial Chemoembolization Alone in Patients with Unresectable Hepatocellular Carcinoma. Liver Cancer. 2022 Feb 10;11(4):354-367. doi: 10.1159/000522547. eCollection 2022 Jul. PMID 35978604
- [Derived] Kudo M, Ueshima K, Ikeda M, Torimura T, Tanabe N, Aikata H, Izumi N, Yamasaki T, Nojiri S, Hino K, Tsumura H, Kuzuya T, Isoda N, Yasui K, Aino H, Ido A, Kawabe N, Nakao K, Wada Y, Yokosuka O, Yoshimura K, Okusaka T, Furuse J, Kokudo N, Okita K, Johnson PJ, Arai Y; TACTICS study group. Randomised, multicentre prospective trial of transarterial chemoembolisation (TACE) plus sorafenib as compared with TACE alone in patients with hepatocellular carcinoma: TACTICS trial. Gut. 2020 Aug;69(8):1492-1501. doi: 10.1136/gutjnl-2019-318934. Epub 2019 Dec 4. PMID 31801872